CLINICAL TRIAL: NCT02791087
Title: Investigation of the Role of Hemodynamics in Re-stenosis of CABG Patients
Status: Completed | Type: Observational
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/366/C
Record Dates: First submitted 2016-05-31; First posted 2016-06-06 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2017-09

CONDITIONS: Coronary Artery Disease; Stable Angina; Unstable Angina
MeSH Terms: conditions — Coronary Artery Disease; Angina, Stable; Angina, Unstable

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Coronary Artery Disease for CABG: Patients undergoing or underwent Coronary Bypass Surgery with at least one saphenous vein graft. Intra-operative graft flow rate measurement will be done during CABG surgery.
  Interventions: Other: Computed Tomography Angiography; Other: Intra-operative graft flow rate measurement
- Stable/Unstable Angina: Patients with no known history of coronary artery disease undergoing Computed Tomography Angiography scan due to stable/Unstable Angina.
  Interventions: Other: Computed Tomography Angiography

INTERVENTIONS:
Other: Computed Tomography Angiography — The CTA is non-invasive and is used commonly for patients who have chest pain to assess the coronary artery disease, prior to the more invasive coronary angiogram.
Other: Intra-operative graft flow rate measurement — This procedure involves the insertion of a Medistim Ultrasound Transit Time Flow Probe into the graft vessel to measure its flow rate. This technique is commonly used for evaluating graft opening during CABG surgery.
  Groups: Coronary Artery Disease for CABG

SUMMARY:
CFD simulations in this study provide detailed hemodynamics information, which cannot be obtained from cardiac images alone. The investigators hypothesize that our proposed simulations will provide strong correlation between hemodynamic parameters, such as WSSG and SPA, and clinically identified graft stenosis. These correlations will allow the investigators to identify the future patients at high risk of graft stenosis and lead to future researches on optimizing and refining surgical plans, such as finding optimal proximal and distal anastomoses locations, optimal graft length and diameter, which could lead to improved longevity of the graft. Once CFD coupled shape optimizer is validated, it could be part of the surgical simulator to help in training the next generation physicians. It could provide new viewpoints for assessing whether some modified surgical techniques are better or not. It could also aid in designing and evaluating the vascular medical devices, including stent, artificial graft, and etc., which would lead to better surgical outcome.

DETAILED DESCRIPTION:
Since the introduction of saphenous vein grafting in the late 1960s, CABG, with or without arterial conduits, remains the gold standard for management of intractable angina due to coronary artery occlusive disease. According to the statistics of American Heart Association, 571,000 of bypass procedures were performed on 355,000 patients in 1999. In Singapore, 831 CABG surgeries were carried out in 2011. With the aging of society, the number of bypass operations is suspected to keep increasing over the years.

However, the CABG was not without complications. The saphenous vein, which is the most commonly used vessel for grafting, provides only palliation of the ongoing process. Approximately 15% to 20% saphenous vein grafts occlude in the first year. An additional 2% to 5% grafts occlude each year between 2 to 10 years postoperatively. At 10 to 14 years, 50% of the grafts are occluded. Similar data is reported in 2011 ACCF/AHA CABG guideline. Although thrombosis, intimal hyperplasia and atherosclerosis are found by pathological examinations, the exact mechanism of stenosis is still not fully understood. The investigators hypothesize that localized hemodynamic parameters is related to the sites of graft occlusion.

Hemodynamic parameters are propounded to be involved in localization of arterial stenosis in literatures. High wall shear stress was found to lead abnormal endothelia cells by Fry on the study of thoracic aorta in dogs. Intimal thicken and atherosclerosis was found to be developed in the low WSS region when studying stenosis on postmortem human carotid bifurcations, synthetic grafts on dog's carotid arteries and human coronary arteries. Both high and low WSS segments was found to interplay with plaque development on human coronary arteries. Bovine aortic endothelial cells density was found to increase in the high wall shear stress gradient regions by Depaola and colleagues. Significantly increased WSSG was found at the throat of the cervical carotid stenosis by Schirmer and colleagues for 8 patients. Stress phase angle was proposed to be a useful indicator in predicting sites prone to atherosclerosis by Torii et al. when investigating a patient's right coronary artery with stenosis. Low-density lipoprotein transportation was proposed to be a useful indicator in predicting sites prone to atherosclerosis on human left coronary artery by Olgac and colleagues.

All of these hemodynamic parameters are related to the forces acting on the endocellar cells, especially the wall shear stress. Signaling pathways have been proposed, which mediate the mechano- chemical transduction in endothelial cells in response to disturbed WSS. Among the WSS-related parameters, WSSG and SPA may be the most important, as WSSG measures the impact of changes in surface forces, while SPA refers to the phase angle between WSS and WCS. Therefore direct study on the human with CABG is necessary to provide strong correlation between graft stenosis and hemodynamic parameters, which would be helpful in identifying the patients at high risk of re-stenosis and optimizing the surgery from a mechanical standpoint. The current project aims to fill in this gap.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-80.
* Undergoing or underwent CABG with at least one saphenous vein graft. (Only for recruitment of CABG patients)
* No known history of coronary artery disease (only for recruitment of volunteers with Stable/unstable angina).

Exclusion Criteria:

* Individuals unable to provide informed consent.
* Non-cardiac illness with life expectancy <2 years.
* Pregnant state.
* Allergy to iodinated contrast.
* Significant arrhythmia; heart rate ≥ 100 beats/min; systolic blood pressure ≤90 mmHg.
* Renal dysfunction(Glomerular filtration rate (GFR) <30 mL/min/1.73m2).
* Contraindication to beta blockers or nitroglycerin.
* Canadian Cardiovascular Society class IV angina.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential patients scheduled for Coronary Bypass Surgery identified at NHCS cardiology inpatient and patients with stable/unstable angina from cardiology inpatient and outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2013-06; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Evidence of allergic reaction due to CTA scan contrast | Within first day after scan

CONTACTS AND LOCATIONS:
Overall Officials: Junmei Zhang, Principal Investigator — National Heart Centre Singapore
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No